CLINICAL TRIAL: NCT02748772
Title: Application of Two Anti-angiogenesis Drugs Combined With Chemotherapy in Advanced Colorectal Cancer Under the Background of Precision Medical
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First People's Hospital of Hefei (Other)
Collaborators: Anhui Provincial Cancer Hospital (Other); Anhui Jimin Cancer Hospital (Unknown); Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FirstPeoplesHHeFei
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Neoplasms
Keywords: Anti-angiogenesis Drugs; Advanced Colorectal Cancer; Endostar; Thalidomide; Vascular Endothelial Growth Factor A
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two Anti-angiogenesis Drugs（Endostar and Thalidomide） (Active Comparator): Two Anti-angiogenesis Drugs（Endostar and Thalidomide） Combined With Chemotherapy for the patients of Advanced Colorectal Cancer
  Interventions: Drug: Two Anti-angiogenesis Drugs（Endostar and Thalidomide）; Drug: Pure chemotherapy（Xelox）
- Pure chemotherapy（Xelox） (Placebo Comparator): chemotherapy alone for the patients of Advanced Colorectal Cancer
  Interventions: Drug: Pure chemotherapy（Xelox）

INTERVENTIONS:
Drug: Two Anti-angiogenesis Drugs（Endostar and Thalidomide） — Endostar:30 mg/d, CIV (continous intravenous pumping) on day 7 of each 21 day cycle，5 days before the chemotherapy is the first day; Thalidomide:100-200mg/d,PO (peros) on day 14 of each 21 day cycle Number of Cycles: 6 cycle or progression or unacceptable toxicity develops.
  Other Names: rh-Endostatin；Distaval
  Arms: Two Anti-angiogenesis Drugs（Endostar and Thalidomide）
Drug: Pure chemotherapy（Xelox） — CapeOX (also called XELOX) is a chemotherapy regimen consisting of capecitabine (trade name Xeloda) combined with oxaliplatin.
  Oxaliplatin 130mg/m2 IV over 2 hours,day1 Capecitabine 850-1000mg/m2 twice daily PO for 14 days Repeat every 3 weeks Number of Cycles: 6 cycle or progression or unacceptable toxicity develops.
  Other Names: CapeOX

SUMMARY:
The purpose of this study is to determine whether Endostar pumping into vein with Thalidomide are more effective in the treatment of Advanced Colorectal Cancer (ACRC).

DETAILED DESCRIPTION:
Endostar have anti-tumor activity by against vascular endothelial growth factor.

Thalidomide is a therapeutic for insomnia and vomiting. It is also used for tumor treatment as an Anti-angiogenesis drug and immune regulator in recently years.

1. Evaluated the therapeutic effects and survival benefits of ACRC treatment by using the Endostar and Thalidomide combined with XELOX regimens. (including the RR, DCR, PFS, and QOL);
2. Evaluated the security and tolerance by treating with Endostar and Thalidomide (the occurrence of adverse reaction, the degree, the regularity and control measures, etc.);
3. Detected the histological markers (VEGF/VEGFR, PDGF/PDGFR, BFGF/FGFR, cox-2, Her-2, K-Ras and p53) before the patients into the group. Make a retrospective analysis of individual molecules indicators to guide significant therapy of ACRC.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with stage IV colorectal cancer can't receive operative treatment diagnosed by Histopathological or cytological examination or can receive operation after conversion therapy.
2. The niave patients relapse and metastasize after more than 6 months' chemotherapeutic diapause after operation or adjuvant chemotherapy or refuse to another operate or need operate only after conversion therapy
3. Have at least one measurable nidus, Ordinary CT or MRI scan nidus 20 mm or higher, Spiral CT and PET - CT scan nidus 10 mm or higher.
4. The first 3 weeks before entering the group have stopped chemotherapy or radiotherapy and recovered from previous treatment of toxic effects. The patients who have received the treatment of delayed toxicity drugs (such as mitomycin or nitrourea) should stop treatment of 6 weeks;
5. ECOG score of 0 to 2 points.
6. Expected survival period for 3 months or more.
7. Aged 18 to 75 years of age, and gender not limited.
8. The electrocardiogram is normal and the body doesn't have unhealed wounds.
9. Peripheral blood cell count, WBC 4.0 x 109 / L or higher, PLT 80 x 109 / L or higher, Hb 90 g/L or higher.
10. Renal function, Cr 2.0 x UNL (upper limit of normal) or less.
11. Liver function, AST, ALT were 2.5 times the normal limit or less (if identified as liver metastasis, five times the normal limit or less).
12. Previous have no severe allergic reactions on biological agents, especially e. coli genetically engineered products.
13. Voluntary to participate in groups, good compliance, willing to cooperate with test observation and sign a written informed consent.

Exclusion Criteria:

1. Pregnant, lactating women,or female patient who have fertility ability but have not taken contraceptive measures;
2. Patients who exist serious acute infection and have not been controlled；or patients who exist purulent infection,chronic infection and delayed wound healing;
3. Patients with serious heart disease, including:congestive heart failure ,uncontrollable high-risk arrhythmias,unstable angina, myocardial infarction, severe heart valve disease and resistant hypertension;
4. Patients whose target lesions had previously received radiation therapy or other topical treatment(radio frequency, ultrasonic, freezing);
5. Patients who suffered from uncontrollable neurological and psychiatric diseases or mental disorders, have poor compliance as well as can not cope with others and failed to narrative therapy respond;patients whose primary brain or central nervous system metastases disease had not been controlled and those with Cranial hypertension or neuropsychiatric symptoms;
6. Patients who had meanwhile participated in other clinical trials;
7. Other circumstances which researchers considered that patients should not participate in this test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 Years
  Adoption of internationally accepted evaluation oncology research progression-free survival (PFS) as a main observation indexes.

SECONDARY OUTCOMES:
RR | 2 Years
  Response Evaluation Criteria In Solid Tumors (RECIST) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment. divided into complete remission (CR), partial response (PR), stable (SD) and development (PD). The total effective rate (RR) refers to the percentage of CR + PR.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Anhui Cancer Hospital, Hefei, Anhui
  - Anhui Jimin Cancer Hospital, Hefei, Anhui
  - The First People's Hospital of Hefei, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gamelin E, Delva R, Jacob J, Merrouche Y, Raoul JL, Pezet D, Dorval E, Piot G, Morel A, Boisdron-Celle M. Individual fluorouracil dose adjustment based on pharmacokinetic follow-up compared with conventional dosage: results of a multicenter randomized trial of patients with metastatic colorectal cancer. J Clin Oncol. 2008 May 1;26(13):2099-105. doi: 10.1200/JCO.2007.13.3934. PMID 18445839
- [Background] Haller DG, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Gilberg F, Rittweger K, Schmoll HJ. Capecitabine plus oxaliplatin compared with fluorouracil and folinic acid as adjuvant therapy for stage III colon cancer. J Clin Oncol. 2011 Apr 10;29(11):1465-71. doi: 10.1200/JCO.2010.33.6297. Epub 2011 Mar 7. PMID 21383294
- [Background] Folkman J. Angiogenesis: an organizing principle for drug discovery? Nat Rev Drug Discov. 2007 Apr;6(4):273-86. doi: 10.1038/nrd2115. PMID 17396134
- [Background] O'Reilly MS, Boehm T, Shing Y, Fukai N, Vasios G, Lane WS, Flynn E, Birkhead JR, Olsen BR, Folkman J. Endostatin: an endogenous inhibitor of angiogenesis and tumor growth. Cell. 1997 Jan 24;88(2):277-85. doi: 10.1016/s0092-8674(00)81848-6. PMID 9008168
- [Background] Wang J, Sun Y, Liu Y, Yu Q, Zhang Y, Li K, Zhu Y, Zhou Q, Hou M, Guan Z, Li W, Zhuang W, Wang D, Liang H, Qin F, Lu H, Liu X, Sun H, Zhang Y, Wang J, Luo S, Yang R, Tu Y, Wang X, Song S, Zhou J, You L, Wang J, Yao C. [Results of randomized, multicenter, double-blind phase III trial of rh-endostatin (YH-16) in treatment of advanced non-small cell lung cancer patients]. Zhongguo Fei Ai Za Zhi. 2005 Aug 20;8(4):283-90. doi: 10.3779/j.issn.1009-3419.2005.04.07. Chinese. PMID 21108883
- [Background] Ling Y, Yang Y, Lu N, You QD, Wang S, Gao Y, Chen Y, Guo QL. Endostar, a novel recombinant human endostatin, exerts antiangiogenic effect via blocking VEGF-induced tyrosine phosphorylation of KDR/Flk-1 of endothelial cells. Biochem Biophys Res Commun. 2007 Sep 14;361(1):79-84. doi: 10.1016/j.bbrc.2007.06.155. Epub 2007 Jul 10. PMID 17644065
- [Background] Kim YM, Hwang S, Kim YM, Pyun BJ, Kim TY, Lee ST, Gho YS, Kwon YG. Endostatin blocks vascular endothelial growth factor-mediated signaling via direct interaction with KDR/Flk-1. J Biol Chem. 2002 Aug 2;277(31):27872-9. doi: 10.1074/jbc.M202771200. Epub 2002 May 23. PMID 12029087
- [Background] Li XQ, Shang BY, Wang DC, Zhang SH, Wu SY, Zhen YS. Endostar, a modified recombinant human endostatin, exhibits synergistic effects with dexamethasone on angiogenesis and hepatoma growth. Cancer Lett. 2011 Feb 28;301(2):212-20. doi: 10.1016/j.canlet.2010.12.004. Epub 2011 Jan 7. PMID 21216091
- [Background] Dahut WL, Gulley JL, Arlen PM, Liu Y, Fedenko KM, Steinberg SM, Wright JJ, Parnes H, Chen CC, Jones E, Parker CE, Linehan WM, Figg WD. Randomized phase II trial of docetaxel plus thalidomide in androgen-independent prostate cancer. J Clin Oncol. 2004 Jul 1;22(13):2532-9. doi: 10.1200/JCO.2004.05.074. PMID 15226321
- [Background] McMeekin DS, Sill MW, Darcy KM, Stearns-Kurosawa DJ, Webster K, Waggoner S, Benbrook D. A phase II trial of thalidomide in patients with refractory leiomyosarcoma of the uterus and correlation with biomarkers of angiogenesis: a gynecologic oncology group study. Gynecol Oncol. 2007 Sep;106(3):596-603. doi: 10.1016/j.ygyno.2007.05.013. Epub 2007 Jun 27. PMID 17597196
- [Background] Dredge K, Marriott JB, Macdonald CD, Man HW, Chen R, Muller GW, Stirling D, Dalgleish AG. Novel thalidomide analogues display anti-angiogenic activity independently of immunomodulatory effects. Br J Cancer. 2002 Nov 4;87(10):1166-72. doi: 10.1038/sj.bjc.6600607. PMID 12402158
- [Background] Gupta D, Treon SP, Shima Y, Hideshima T, Podar K, Tai YT, Lin B, Lentzsch S, Davies FE, Chauhan D, Schlossman RL, Richardson P, Ralph P, Wu L, Payvandi F, Muller G, Stirling DI, Anderson KC. Adherence of multiple myeloma cells to bone marrow stromal cells upregulates vascular endothelial growth factor secretion: therapeutic applications. Leukemia. 2001 Dec;15(12):1950-61. doi: 10.1038/sj.leu.2402295. PMID 11753617
- [Background] Wang Z, Dabrosin C, Yin X, Fuster MM, Arreola A, Rathmell WK, Generali D, Nagaraju GP, El-Rayes B, Ribatti D, Chen YC, Honoki K, Fujii H, Georgakilas AG, Nowsheen S, Amedei A, Niccolai E, Amin A, Ashraf SS, Helferich B, Yang X, Guha G, Bhakta D, Ciriolo MR, Aquilano K, Chen S, Halicka D, Mohammed SI, Azmi AS, Bilsland A, Keith WN, Jensen LD. Broad targeting of angiogenesis for cancer prevention and therapy. Semin Cancer Biol. 2015 Dec;35 Suppl(Suppl):S224-S243. doi: 10.1016/j.semcancer.2015.01.001. Epub 2015 Jan 16. PMID 25600295
- [Background] Narita K, Fujii T, Ishiwata T, Yamamoto T, Kawamoto Y, Kawahara K, Nakazawa N, Naito Z. Keratinocyte growth factor induces vascular endothelial growth factor-A expression in colorectal cancer cells. Int J Oncol. 2009 Feb;34(2):355-60. PMID 19148469
- [Background] Heldin CH, Westermark B. Mechanism of action and in vivo role of platelet-derived growth factor. Physiol Rev. 1999 Oct;79(4):1283-316. doi: 10.1152/physrev.1999.79.4.1283. PMID 10508235
- [Background] Appelmann I, Liersch R, Kessler T, Mesters RM, Berdel WE. Angiogenesis inhibition in cancer therapy: platelet-derived growth factor (PDGF) and vascular endothelial growth factor (VEGF) and their receptors: biological functions and role in malignancy. Recent Results Cancer Res. 2010;180:51-81. doi: 10.1007/978-3-540-78281-0_5. PMID 20033378
- [Background] Casanovas O, Hicklin DJ, Bergers G, Hanahan D. Drug resistance by evasion of antiangiogenic targeting of VEGF signaling in late-stage pancreatic islet tumors. Cancer Cell. 2005 Oct;8(4):299-309. doi: 10.1016/j.ccr.2005.09.005. PMID 16226705
- [Background] Chao C, Carmical JR, Ives KL, Wood TG, Aronson JF, Gomez GA, Djukom CD, Hellmich MR. CD133+ colon cancer cells are more interactive with the tumor microenvironment than CD133- cells. Lab Invest. 2012 Mar;92(3):420-36. doi: 10.1038/labinvest.2011.185. Epub 2011 Dec 12. PMID 22157717
- [Background] Saukkonen K, Nieminen O, van Rees B, Vilkki S, Harkonen M, Juhola M, Mecklin JP, Sipponen P, Ristimaki A. Expression of cyclooxygenase-2 in dysplasia of the stomach and in intestinal-type gastric adenocarcinoma. Clin Cancer Res. 2001 Jul;7(7):1923-31. PMID 11448905